CLINICAL TRIAL: NCT04434443
Title: Effects of Trunk Exercise on Unstable Surface on Trunk Control and Balance in Persons With Stroke
Brief Title: Effects of Trunk Exercise on Trunk Control and Balance in Persons With Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: Tainan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Principal Investigator, Sang-I Lin, Professor, Department of Physical Therapy, National Cheng Kung University, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-ER-106-428
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cerebrovascular Accident; Balance Impairment
Keywords: stroke; balance; Trunk exercise; Trunk control; standing
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor not aware of group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trunk exercise on unstable surface (Experimental): trunk exercise training in supine and sitting positions, with unstable surfaces
  Interventions: Other: trunk exercise on unstable exercise
- upper limb range of motion exercise (Sham Comparator): upper limb range of motion exercise in sitting with back fully supported
  Interventions: Other: Upper limb range of motion exercise

INTERVENTIONS:
Other: trunk exercise on unstable exercise — Participants would receive exercises on unstable surface. Started from supine position, participants had abdominal drawer-in maneuver with soft foam under the pelvic. Lower trunk rotation, bridging and abdominal muscles isometric contraction exercises were also used in this exercise during supine position, with different unstable surfaces used. Including soft foam under the feet, then progressed to BOSU ball under the feet, then progressed to the a BOSU ball under the feet combined with pelvic on soft foam. During sitting, BOSU ball and Swiss ball were used as unstable surface. Pelvic anterior-posterior tilt, lateral tilting, rotation, lifting, and stepping with arm swing were used in this position.
  Arms: trunk exercise on unstable surface
Other: Upper limb range of motion exercise — Upper limb range of motion exercise with trunk fully supported
  Arms: upper limb range of motion exercise

SUMMARY:
This study examined the effects of trunk exercise on unstable surfaces on trunk control and balance for persons in the sub-acute stage of stroke. The hypothesis was that, compared to upper limb exercises in well supported sitting position, this exercise would lead to better trunk control and sitting and standing balance. The results supported the hypothesis.

DETAILED DESCRIPTION:
Inpatients in the sub-acute stage of stroke were randomly assigned to receive upper limb range of motion exercises in well supported sitting position or trunk exercises on unstable surfaces in supine and sitting, 30 min per session, 2 sessions per week for 6 weeks, in addition to their daily conventional stroke rehabilitation. Sensorimotor functions, including hand grip strength, plantar sensitivity, stroke rehabilitation assessment of movement and Fugl-Meyer lower extremity motor scale, and clinical outcome assessments, including Trunk Impairment Scale and 6-meter walk test, were conducted by a blinded assessor. Biomechanical outcome measures included center of pressure area while maintaining static posture and peak displacement while leaning forward, and the average speed of the unaffected arm raising (to represent the ability to provide a stable foundation for focal movement). These measures were taken in sitting without foot support, sitting with foot support and standing to reflect trunk control, sitting balance and standing balance, respectively.

ELIGIBILITY:
Inclusion Criteria:

* age: between 20-80 years old
* first time stroke
* could sit without back support at least 20 seconds
* could understand and follow experimental instructions

Exclusion Criteria:

* medically unstable
* other neuromuscular/musculoskeletal problems that would affect balance

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Center of pressure | 6 weeks
  range of displacement (cm)
Angular velocity of the non-affected arm raising | 6 weeks
  mean velocity

SECONDARY OUTCOMES:
Trunk Impairment Scale | 6 weeks
  total score (0-23); higher scores mean better outcome
6-meter walking tests | 6 weeks
  time (sec) to walk 6 meters

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan